CLINICAL TRIAL: NCT02823080
Title: Sequential E2 Levels Not Ovarian Maximal Diameter Estimates Were Correlated With Outcome of Cetrotide Therapy for Management of Women at High-risk of Ovarian Hyperstimulation Syndrome
Brief Title: Outcome of Cetrotide Therapy for Management of Women at High-risk of Ovarian Hyperstimulation Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, director clinical research, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Benha U; kmsalama (Registry Identifier: khalid)
Record Dates: First submitted 2016-06-21; First posted 2016-07-06 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — cetrorelix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cetrotide (Active Comparator): study group (24 patients = intervention) received intervention for 3-daysCetrorelix Acetate sc injection (0.25 mg/day) started on Day-0. Serum E2, pain scores and MOD were checked daily. Hematocrit value (Ht%), total leucocytic count (TLC), gastrointestinal (GI) manifestations and ascites grading were re-evaluated on Day-3, 6 and 8.
  Interventions: Drug: Cetrorelix
- no cetrotide (No Intervention): control group (24 patients) did not receive 3-daysCetrorelix Acetate (no intervention). Serum E2, pain scores and MOD were checked daily. Hematocrit value (Ht%), total leucocytic count (TLC), gastrointestinal (GI) manifestations and ascites grading were re-evaluated on Day-3, 6 and 8.

INTERVENTIONS:
Drug: Cetrorelix — study group received 3-day Cetrorelix Acetate sc injection (0.25 mg/day) started on Day-0. Serum E2, pain scores and MOD were checked daily. Hematocrit value (Ht%), total leucocytic count (TLC), gastrointestinal (GI) manifestations and ascites control (24 patients) did not receive Cetrorelix Acetate. Grading were re-evaluated on Day-3, 6 and 8.
  Other Names: cetrotide
  Arms: cetrotide

SUMMARY:
To evaluate safety and efficacy of 3-day cetrotide therapy started on day of oocyte retrieval (Day-0) in women at high-risk for development of ovarian hyperstimulation syndrome (OHSS) after gonadotropin- releasing hormon agonist induction protocol.

Patients & Methods: Forty-eight women fulfilling inclusion criteria underwent ultrasound scanning for maximal ovarian diameter (MOD) estimation and ascites grading. Patients underwent embryo freezing, but study group received 3-day Cetrotide sc injection (0.25 mg/day) started on Day-0. Serum E2, pain scores and MOD were checked daily. Hematocrit value (Ht%), total leucocytic count (TLC), gastrointestinal (GI) manifestations and ascites grading were re-evaluated on Day-3, 6 and 8

DETAILED DESCRIPTION:
The current study is conducted at Assisted Reproduction Unit at Almana general Hospital, kingdom of saudi arabia.and other private centers in Egypt. The study protocol was approved by the Local Ethical Committee. The study aimed to include women suspected to be at high risk for development of OHSS during agonist ovarian stimulation protocol.The study includes only women of couples singed written consent to participate in the study, to undergo embryo freezing and to postpone for transfer of cryopreserved embryo.

All patients are clinically evaluated for the presence of abdominal pain and if present will be graduated using a numerical pain visual analogue scale (VAS) with 0 means no pain and 10 means severe intolerable pain. Patients are evaluated for the presence of nausea and/or vomiting and sense of abdominal distension. Symptoms are scored using verbal analogue scale as nil, mild, moderate, and severe symptom. Blood samples are obtained under complete aseptic condition for estimation of serum E2 level and determination of hematocrit value (Ht%) and total leucocytic count (TLC).

Then, all patients underwent ultrasound scanning for estimation of ovarian measurements that were represented as the maximal ovarian diameter (MOD) and for ascites grading if present. Ultrasound scanning is performed using a 5 megahertz vaginal probe , otherwise a 3.5 megahertz, 2.6 megahertz or 5megahertz abdominal probe is used if visualization using a vaginal probe is compromised. Ascites is graded according to the quantity of fluid accumulation in the peritoneal cavity with the patient in the anti-Trendelenburg position.

Women fulfilling inclusion criteria were randomely allocated,using sealed envelops, into two equal groups. Group with embryo freezing alone (Control group) or while the other group additionally receives cetrotide subcutaneous injection in a daily dose of 0.25 mg started on day of oocyte retrieval for 3 days (Study group). Symptomatic treatment for associated symptoms as analgesics, antiemetics and antispasmodics are also prescribed. Patients are categorized according to classification grading of OHSS.

Class Clinical features Biochemical features

Mild - Abdominal distension/ discomfort

* Mild nausea/vomiting
* Diarrhea
* Ovarian size usually < 8 cm No clinically important laboratory findings

Moderate - Mild features plus

* US evidence of ascites - Elevated Ht (>41%)
* Elevated TLC >15,000/ ml
* Hypoproteinemia

Severe - Mild & Moderate features plus

* Clinically detected ascites
* Severe abdominal pain
* Intractable nausea
* Rapid weight gain (>1 kg/24 hr)
* Pleural effusion
* Severe dyspnea
* Oliguria/anuria
* Low blood/central venous pressures
* Syncope
* Venous thrombosis
* Hemoconcentration (Ht >55%)
* TLC >25,000/ ml
* Serum creatinine >1.6 mg/dl
* creatinine clearance <50 ml/min
* Hyponatremia (Na+<135milliequivalent per litre)
* Hypokalemia (K+ < 5 milliequivalent per litre)
* Elevated liver enzymes

Critical - Severe features plus

* Anuria/ Acute renal failure
* Arrhythmia
* Pericardial effusion
* Massive hydrothorax
* Thrombo-embolism
* Arterial thrombosis
* (ARDS)Adult respiratory distress syndrome
* Sepsis - Worsening of biochemical

findings seen with severe OHSS

US: Ultrasound; Ht%:Ht; Hematocrit value; TLC: Total leucocytic count: ARDS; adult respiratory distress syndrome.

All patients are managed as outpatients unless management of severe symptoms necessitated hospital admission. Pain scores, serum E2 levels and MOD are evaluated daily. Patients are evaluated for associated symptoms previously determined during clinical evaluation, ascites grading and TLC and Ht value were evaluated at 3 and 6 days and on end of the trial on the 8th day after oocyte retrieval.

ELIGIBILITY:
Inclusion Criteria:

1. number of retrieved oocytes was ≥20
2. mean number of follicles with a diameter of >16 mm was ≥18
3. serum E2 concentrations of ≥3500 pg/ml
4. ovarian diameter on the day of ovum retrieval of >10 cm
5. presentation of evident symptoms of OHSS on the day of aspiration .

Exclusion Criteria:

1- Absence of one or more of the items of the inclusion criteria.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: khalid M salama, MD, Principal Investigator — Benha University
Locations (1):
- Benha university hospitalا, Banhā, El Qalubia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Lainas TG, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas GT, Kolibianakis EM. Management of severe early ovarian hyperstimulation syndrome by re-initiation of GnRH antagonist. Reprod Biomed Online. 2007 Oct;15(4):408-12. doi: 10.1016/s1472-6483(10)60366-5. PMID 17908403
- [Background] Albano C, Smitz J, Camus M, Riethmuller-Winzen H, Van Steirteghem A, Devroey P. Comparison of different doses of gonadotropin-releasing hormone antagonist Cetrorelix during controlled ovarian hyperstimulation. Fertil Steril. 1997 May;67(5):917-22. doi: 10.1016/s0015-0282(97)81407-0. PMID 9130900
- [Background] Navot D, Bergh PA, Laufer N. Ovarian hyperstimulation syndrome in novel reproductive technologies: prevention and treatment. Fertil Steril. 1992 Aug;58(2):249-61. doi: 10.1016/s0015-0282(16)55188-7. PMID 1633889
- [Derived] Salama KM, Abo Ragab HM, El Sherbiny MF, Morsi AA, Souidan II. Sequential E2 levels not ovarian maximal diameter estimates were correlated with outcome of cetrotide therapy for management of women at high-risk of ovarian hyperstimulation syndrome: a randomized controlled study. BMC Womens Health. 2017 Nov 13;17(1):108. doi: 10.1186/s12905-017-0466-z. PMID 29132339
- See also: infertility — http://bu.edu.eg

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetrotide: study group (24 patients = intervention) received intervention for 3-daysCetrorelix Acetate sc injection (0.25 mg/day) started on Day-0. Serum E2, pain scores and MOD(maximal ovarian diameter) were checked daily. Hematocrit value (Ht%), total leucocytic count (TLC), gastrointestinal (GI) manifestations and ascites grading were re-evaluated on Day-3, 6 and 8.
Period: Overall Study
Arm/Group | Cetrotide | no Cetrotide
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetrotide | no Cetrotide | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 12 | 12 | 24
  Saudi Arabia | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Daily Serum E2 Levels
Description: Serum E2 levels (Serum E2 level in picograms/ml) were evaluated daily.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: picograms/ml
Arm/Group | Cetrotide | no Cetrotide
Number analyzed (Participants) | 24 | 24
picograms/ml
  Day-0 | 4761 (940) | 5004 (792)
  Day-1 | 3397 (1361) | 4212 (950)
  Day-2 | 2772 (1456) | 3620 (1037)
  Day-3 | 2067 (900) | 3592 (862)
  Day-4 | 1452 (617) | 2570 (914)
  Day-5 | 1173 (180) | 1914 (965)
  Day-6 | 1173 (180) | 1544 (812)
  Day-7 | 969 (118) | 1275 (588)
  Day-8 | 902 (66) | 1044 (200)
Statistical Analysis 1: Comparison: Cetrotide vs no Cetrotide; Test type: Other; p < 0.05, ANOVA

2. Primary Outcome: Daily Maximal Ovarian Diameter
Description: MOD (maximal ovarian diameter in mm) were evaluated daily.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cetrotide | no Cetrotide
Number analyzed (Participants) | 24 | 24
mm
  Day-0 | 9.4 (4.5) | 10.4 (5.8)
  Day-1 | 9.3 (4.6) | 10.2 (5.6)
  Day-2 | 9.1 (4.2) | 9.6 (4.6)
  Day-3 | 8.7 (4.3) | 9.4 (4.9)
  Day-4 | 8.5 (4.3) | 9.2 (4.7)
  Day-5 | 7.8 (4) | 9 (4.6)
  Day-6 | 7.5 (4.2) | 8.5 (4.6)
  Day-7 | 7.3 (4) | 8.2 (4.5)
  Day-8 | 7.1 (3.7) | 7.9 (4.2)
Statistical Analysis 1: Comparison: Cetrotide vs no Cetrotide; Test type: Other; p < 0.05, ANOVA

3. Secondary Outcome: Daily Numerical Pain Visual Analogue Scale Score
Description: -All patients were clinically evaluated for the presence of abdominal pain and if present was graduated using a numerical pain visual analogue scale (VAS) with 0 means no pain and 10 means severe intolerable pain .
Time Frame: 8 days.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cetrotide: study group (24 patients = intervention) received intervention for 3-days Cetrorelix Acetate sc injection (0.25 mg/day) started on Day-0. Serum E2, pain scores and MOD were checked daily. Hematocrit value (Ht%), total leucocytic count (TLC), gastrointestinal (GI) manifestations and ascites grading were re-evaluated on Day-3, 6 and 8.
Arm/Group | Cetrotide | no Cetrotide
Number analyzed (Participants) | 24 | 24
units on a scale
  Day-0 | 5.3 (1.6) | 5.4 (1.7)
  Day-1 | 4.3 (1.3) | 5 (1.3)
  Day-2 | 3.6 (1) | 4.9 (1.8)
  Day-3 | 2.3 (1.8) | 4.6 (1.8)
  Day-4 | 1.6 (1.2) | 4.5 (1.4)
  Day-5 | 0.92 (1.1) | 3.7 (2)
  Day-6 | 0.33 (0.6) | 2.4 (1.1)
  Day-7 | 0.17 (0.38) | 1.6 (1.1)
  Day-8 | 0.13 (0.34) | 1.1 (1.7)
Statistical Analysis 1: Comparison: Cetrotide vs no Cetrotide; Test type: Other; p < 0.05, ANOVA

4. Secondary Outcome: Daily Hematocrits Value
Description: Blood samples were obtained under complete aseptic condition for determination of hematocrits value (Ht%)
Time Frame: 0-8 days.
Measure: Mean (Standard Deviation); unit: percentge
Arm/Group | Cetrotide | no Cetrotide
Number analyzed (Participants) | 24 | 24
percentge
  Day-0 | 42.2 (5.2) | 39.8 (4.2)
  Day-3 | 38.7 (3.3) | 38.8 (3.3)
  Day-6 | 37.3 (2.5) | 38 (3.1)
  Day-8 | 36.8 (2.6) | 37.5 (1.5)

5. Secondary Outcome: Ultrasound Detected Severity Grades of Ascites From Days 0-8
Description: -US detected severity grades of ascites determined at Day -0, Day -3 and Day -8.
Time Frame: 0-8 days
Measure: Number; unit: US detected ascitis
Arm/Group | Cetrotide | no Cetrotide
Number analyzed (Participants) | 24 | 24
US detected ascitis
  Low grade ascitis at Day-0 | 8 | 6
  Low grade ascitis at Day-3 | 18 | 13
  Low grade ascitis at Day-8 | 21 | 17
  moderate grade ascitis at Day-0 | 16 | 18
  moderate grade ascitis at Day-3 | 6 | 8
  moderate grade ascitis at Day-8 | 3 | 5
  severe grade ascitis at Day-0 | 0 | 0
  severe grade ascitis at Day-3 | 0 | 3
  severe grade ascitis at Day-8 | 0 | 2

6. Secondary Outcome: Daily Total Leucocytic Count
Description: TLC(x 1ooo cells/ml)
Time Frame: 0 -8days.
Measure: Mean (Standard Deviation); unit: 1000 cells/ml
Arm/Group | Cetrotide | no Cetrotide
Number analyzed (Participants) | 24 | 24
1000 cells/ml
  Day-0 | 12.75 (3.1) | 11.6 (3.7)
  Day-3 | 11.5 (2.8) | 11.3 (3.6)
  Day-6 | 11 (1.9) | 11.2 (3.6)
  Day-8 | 9.75 (3.1) | 10.1 (2.2)

7. Other Pre Specified Outcome: Resolution of Gastrointestinal Manifestations Determined Prior to Start of Therapy
Description: -severity grades of gastrointestinal manifestations determined at Day -0,Day -3 and Day -6.
Time Frame: 0-6 days
Measure: Number; unit: GI manifestations
Arm/Group | Cetrotide | no Cetrotide
Number analyzed (Participants) | 24 | 24
GI manifestations
  Nil Nausea at Day-0 | 5 | 6
  mild Nausea at Day-0 | 8 | 7
  moderate Nausea at Day-0 | 7 | 6
  severe Nausea at Day-0 | 4 | 5
  Nil Nausea at Day-3 | 19 | 12
  mild Nausea at Day-3 | 4 | 8
  moderate Nausea at Day-3 | 1 | 4
  severe Nausea at Day-3 | 0 | 0
  Nil Nausea at Day-6 | 24 | 22
  mild Nausea at Day-6 | 0 | 2
  moderate Nausea at Day-6 | 0 | 0
  severe Nausea at Day-6 | 0 | 0
  Nil Vomiting at Day-0 | 14 | 12
  mild Vomiting at Day-0 | 7 | 8
  moderatel Vomiting at Day-0 | 2 | 4
  severe Vomiting at Day-0 | 1 | 0
  Nil Vomiting at Day-3 | 24 | 20
  mild Vomiting at Day-3 | 0 | 4
  moderate Vomiting at Day-3 | 0 | 0
  severe Vomiting at Day-3 | 0 | 0
  Nil Vomiting at Day-6 | 24 | 24
  mild Vomiting at Day-6 | 0 | 0
  moderat Vomiting at Day-6 | 0 | 0
  severe Vomiting at Day-6 | 0 | 0
  Nil Abdominal distension at Day-0 | 5 | 4
  mild Abdominal distension at Day-0 | 8 | 7
  moderate Abdominal distension at Day-0 | 9 | 10
  severe Abdominal distension at Day-0 | 2 | 3
  Nil Abdominal distension at Day-3 | 15 | 9
  mild Abdominal distension at Day-3 | 8 | 12
  moderate Abdominal distension at Day-3 | 1 | 3
  severe Abdominal distension at Day-3 | 0 | 0
  Nil Abdominal distension at Day-6 | 24 | 20
  mild Abdominal distension at Day-6 | 0 | 4
  moderate Abdominal distension at Day-6 | 0 | 0
  severe Abdominal distension at Day-6 | 0 | 0
Statistical Analysis 1: Comparison: Cetrotide vs no Cetrotide; Test type: Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | Cetrotide | no Cetrotide
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
no Limitations and Caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes